CLINICAL TRIAL: NCT07102875
Title: Pilot Study "Ready to Sail 2": Evaluation of the Feasibility and Safety of Sail-Assisted Telerehabilitation in Patients With Rare Skeletal Diseases - Assessment of Motor, Psychosocial, and Quality of Life Outcomes
Brief Title: Ready to Sail 2: A Pilot Study of Sail-Assisted Telerehabilitation in Rare Skeletal Diseases
Acronym: PaS2-EXTEND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Luca Sangiorgi, Director of Rare Skeletal Disorders Department, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 363/2025/Sper/IOR
Record Dates: First submitted 2025-07-14; First posted 2025-08-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Rare Bone Disorders
Keywords: Rare Diseases; Musculoskeletal Diseases; Telerehabilitation; Physical Therapy Modalities; Games, Recreational; Quality of Life; Feasibility Study; Social Behavior; Psychological Well-Being; Adolescent; Young Adult; Wearable Devices; Biomechanical Movement Capture
MeSH Terms: conditions — Rare Diseases; Musculoskeletal Diseases; Social Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sailing Intervention Followed by Home-Based Telerehabilitation Program (Experimental): Participants assigned to this arm will receive a 5-day intensive sailing intervention program, followed by a 3-month home-based telerehabilitation program. The sailing includes daily group-based sailing activities and debriefing activities aimed at enhancing motor skills, coordination, and psychosocial well-being. After the sailing phase, participants will engage in remote physical therapy sessions twice a week via a supervised digital platform. The telerehabilitation component includes progressive exercises targeting balance, proprioception, and functional strength.
  Interventions: Behavioral: Sailing Intervention Plus Home-Based Telerehabilitation
- Home-Based Telerehabilitation Program (Active Comparator): Participants in this arm will undergo a 3-month home-based telerehabilitation program. The intervention consists of two weekly remote sessions conducted via an accredited digital platform. Each session includes warm-up, structured motor and postural exercises, and cool-down/stretching phases. Exercises are progressive and tailored to individual functional capacities, with the goal of improving balance, coordination, and physical function. No sailing therapy is included in this arm.
  Interventions: Behavioral: Home-Based Telerehabilitation

INTERVENTIONS:
Behavioral: Sailing Intervention Plus Home-Based Telerehabilitation — A two-phase rehabilitation program combining 5 days of intensive sailing therapy with a 3-month home-based telerehabilitation plan. The sailing component includes group-based activities in adapted sailing environments, conducted in Marina di Ravenna or Palermo, with daily debriefing and psychosocial support. The telerehabilitation component includes twice-weekly supervised sessions delivered via a digital platform, focusing on progressive motor, proprioceptive, and postural exercises. The intervention aims to improve motor function, quality of life, and psychosocial well-being in individuals with rare skeletal disorders.
  Other Names: 5-day sailing activity
  Arms: Sailing Intervention Followed by Home-Based Telerehabilitation Program
Behavioral: Home-Based Telerehabilitation — Participants perform a 3-month home-based rehabilitation program consisting of two remote sessions per week via a supervised digital platform. Each session includes warm-up, strength and coordination exercises, and cool-down. Exercises are progressive and standardized, but adapted to individual needs to ensure safety and adherence. The intervention targets motor function, balance, proprioception, and psychosocial outcomes, without any sailing component. This arm serves as the active comparator.
  Arms: Home-Based Telerehabilitation Program

SUMMARY:
"Ready to Sail 2 - EXTEND" is a pilot randomized interventional trial designed to assess the feasibility, safety, and preliminary impact of an innovative rehabilitation model combining sailing therapy (velatherapy) with a remote telerehabilitation maintenance program in young individuals with rare skeletal disorders. Building on the promising results of the previous Ready to Sail feasibility study (NCT06397443), this study aims to validate and compare two rehabilitative approaches.

A total of 24 patients aged 12-30 years with a confirmed diagnosis of a rare skeletal disorder will be randomly assigned (1:1) to either:

* Group 1 (Experimental): a 5-day intensive sailing therapy intervention followed by a 3-month personalized telerehabilitation program at home; or
* Group 2 (Active Control): a 3-month telerehabilitation-only program with identical frequency and progression.

The primary objective is to evaluate the feasibility of the experimental program, in terms of adherence, acceptability, and safety. Secondary outcomes include motor functionality (measured by inertial sensors), psychosocial well-being (assessed through validated PROMs), health-related quality of life, and pain perception. The study also explores the medium-term sustainability of rehabilitation outcomes and the influence of individual variables (e.g., age, gender, disease subtype).

The intervention is delivered through a multidisciplinary, patient-centered approach involving rare disease experts, physiatrists, biomechanical engineers, and partner sailing organizations. Sail training activities are adapted for safety and inclusion, and are conducted in two coastal settings (Marina di Ravenna and Palermo), ensuring geographical balance for participant accessibility.

This trial seeks to strengthen the evidence base for integrated, inclusive, and scalable rehabilitation models that address both motor and psychosocial dimensions in rare skeletal conditions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 12 to 30 years, of any sex
* Clinical and/or molecular diagnosis of a rare skeletal disorder
* No orthopedic surgery within the past 6 months, unless deemed clinically irrelevant to study participation by the investigator
* Ability to understand and comply with study procedures
* Signed informed consent obtained from the participant or a legal guardian (for minors)

Exclusion Criteria:

* Severe or unstable medical conditions that could interfere with participation (e.g., uncontrolled cardiac or respiratory disease)
* Cognitive or neurological impairments that may hinder adherence to the study protocol
* Participation in similar intensive rehabilitation programs within the past 3 months
* Contraindications to virtual or sailing-based activities, including but not limited to: (a) Severe motion sickness; (b) Vertigo or vestibular disorders; (c) Photosensitive epilepsy
* Musculoskeletal injuries (e.g., fractures or major sprains) occurring within the past 12 months
* Any condition or circumstance that, in the opinion of the investigator, may compromise safety or study compliance
* Decline or inability to provide informed consent

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adherence to Sailing and Home-Based Telerehabilitation | At 6 months after baseline (end of intervention period)
  Defined as the percentage of scheduled sessions completed by each participant. Adherence is considered achieved if ≥75% of scheduled sessions are completed.
  Unit of Measure: Percentage of participants meeting adherence threshold
Acceptability of the Intervention | At 6 months after baseline (end of intervention period)
  Defined by recruitment rate ≥80% and dropout rate <20%. Unit of Measure: Recruitment rate (%), Dropout rate (%)
Safety of the Intervention | At 6 months after baseline (end of intervention period)
  Defined as the absence of serious adverse events related to the intervention. Unit of Measure: Number of participants experiencing a serious adverse event

SECONDARY OUTCOMES:
Change in Motor Function Measured by Inertial Measurement Units | Baseline (T0), up to 1-day after intervention (T1-only for experimental arm), and at 3-Month Follow-Up (T2)
  Motor function will be assessed using wearable inertial measurement units (IMUs) to evaluate postural control, gait parameters, upper limb mobility, and proprioception. Data will be collected through standardized physical tasks and analyzed to detect changes over time.
Change in Health-Related Quality of Life Measured by EQ-5D-5L | Baseline (T0), up to 1-day after intervention (T1-only for experimental arm), and at 3-Month Follow-Up (T2)
  Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. This instrument includes:
  1. EQ-5D-5L Index Value, ranging from -0.232 to 1.000 (where 1.000 indicates full health, 0 indicates death-equivalent health, and negative values represent health states considered worse than death; higher scores indicate better health status).
  2. EQ Visual Analog Scale (EQ-VAS), ranging from 0 to 100, where 0 represents the "worst imaginable health state" and 100 represents the "best imaginable health state." Higher scores indicate better self-rated health.
  Unit of Measure: EQ-5D-5L Index Value (-0.281 to 1.000); EQ-VAS Score (0 to 100)
Change in Psychosocial Functioning Measured by BESSI-45 | Baseline (T0), up to 1-day after intervention (T1-only for experimental arm), and at 3-Month Follow-Up (T2)
  Psychosocial functioning will be assessed using the Behavioral, Emotional, and Social Skills Inventory (BESSI-45). The BESSI-45 includes 45 items rated on a 5-point Likert scale (1 = "Not at all well" to 5 = "Extremely well"), covering five domains: Self-Management, Social Engagement, Cooperation, Emotional Resilience, and Innovation Skills. Total scores range from 45 to 225, with higher scores reflecting greater psychosocial skills and better psychosocial functioning.
  Unit of Measure: BESSI-45 total score (range 45-225)
Change in Functional Outcomes Measured by PODCI | Baseline (T0), up to 1-day after intervention (T1-only for experimental arm), and at 3-Month Follow-Up (T2)
  Functional health outcomes will be assessed using the Pediatric Outcomes Data Collection Instrument (PODCI), which includes domains such as upper extremity function, mobility, sports and physical activity, pain, happiness, and global function.
Change in Pain Intensity Measured by Visual Analogue Scale (VAS) | Baseline (T0), up to 1-day after intervention (T1-only for experimental arm), and at 3-Month Follow-Up (T2)
  Pain intensity will be assessed using the Visual Analogue Scale for Pain (VAS-Pain), a 10-centimeter horizontal line anchored at the extremes with "0 = no pain" and "10 = worst pain imaginable." Participants mark their current pain level along the line, which is then measured in centimeters from the "no pain" anchor. Scores range from 0 to 10, with higher scores indicating greater pain intensity.
  Unit of Measure: VAS-Pain score (0-10)
Change in Kinesiophobia Measured by Tampa Scale of Kinesiophobia (TSK) | Baseline (T0), up to 1-day after intervention (T1-only for experimental arm), and at 3-Month Follow-Up (T2)
  Fear of movement will be assessed using the Tampa Scale of Kinesiophobia - 13-item version (TSK-13). The TSK-13 includes 13 items rated on a 4-point Likert scale ranging from 1 ("strongly disagree") to 4 ("strongly agree"). Total scores range from 13 to 52, with higher scores indicating greater fear of movement and higher levels of kinesiophobia.
  Unit of Measure: TSK-13 total score (range 13-52)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Boarini M, Romeo A, Banchelli F, Grippa E, Forni S, la Forgia MC, Scognamiglio D, Ferraris PC, Sangiorgi L. Nature-based interventions for individuals with rare skeletal disorders: evaluation of a 5-day sailing program on health-related quality of life. Sci Rep. 2024 Nov 1;14(1):26339. doi: 10.1038/s41598-024-77934-1. PMID 39487306
- [Background] Cappelletti S, Tondo I, Pietrafusa N, Renzetti T, Pannacci I, Gentile S, Perrucci M, Calabrese C, Ferraris PC, Specchio N, Vigevano F. Improvement of quality of life in adolescents with epilepsy after an empowerment and sailing experience. Epilepsy Behav. 2020 May;106:106957. doi: 10.1016/j.yebeh.2020.106957. Epub 2020 Mar 16. PMID 32193096
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- See also: Related Info — https://www.who.int/standards/classifications/international-classification-of-functioning-disability-and-health
- See also: Related Info — https://commission.europa.eu/strategy-and-policy/policies/justice-and-fundamental-rights/disability/union-equality-strategy-rights-persons-disabilities-2021-2030_en
- See also: Related Info — https://partecipa.gov.it/processes/verso-una-piena-inclusione-persone-con-disabilita